CLINICAL TRIAL: NCT07246538
Title: Evaluation of a Novel Positive Airway Pressure System in Volunteers
Brief Title: Positive Airway Pressure (PAP) System Evaluation in Volunteers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Dynasthetics LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB_00190165
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obstruction Airway
Keywords: Device feasibility
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CPAP (Experimental): Airway pressure support through the investigational device
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Airway pressure support through the investigational device.

SUMMARY:
This study will test the control and measurements of a new system for airway support in healthy volunteers. The goals of the study are to evaluate how accurately the system can stabilize airway pressure to a desired level, evaluate the accuracy of the system's reported volume of each breath (tidal volume), evaluate the accuracy of the system's reported respiratory rate, evaluate the accuracy of exhaled carbon dioxide monitoring with a standard carbon dioxide monitor when the novel PAP system is used, and evaluate general comfort of the volunteers while using the system.

DETAILED DESCRIPTION:
Sedation procedures involve administering drugs to patients that reduce awareness and pain without complete loss of consciousness. A common side effect of these drugs is partial or complete obstruction of the airway by the airway tissue, inhibiting the flow of oxygen to the lungs. Research has shown that this risk can be effectively reduced by administering PAP therapy during sedation, which involves directing air flow into a tight-fitting mask over the patient's nostrils and/or mouth. However, non-invasive ventilators used for administering PAP therapy are expensive and large, and often not available in areas of the hospital where sedation procedures take place.

The investigators have developed a small and low-cost novel PAP system for use in sedation procedures that controls airway pressure to desired levels (a feature that is generally only available in larger and higher-cost devices), provides estimates for tidal volumes (generally only available with a non-invasive ventilator), provides respiratory rate estimates, and allows for more accurate monitoring of exhaled carbon dioxide with a standard carbon dioxide monitor using a novel approach that to the investigator's knowledge has not been published. The goal of investigator's study is to demonstrate the accuracy of these features in human subjects. The system is much smaller and less expensive than a non-invasive ventilator, provides enhanced respiratory monitoring, and has the potential to be a practical alternative that would make PAP therapy during sedation much more feasible.

The investigator's evaluation will primarily include evaluating the investigator's system's performance against an FDA cleared commercial respiratory monitor to verify accuracy. The investigators anticipate that the investigator's system will automatically adjust oxygen flow to maintain a desired airway pressure even in the presence of variables such as mask leak and patient inhalation flow. The investigators also anticipate that the investigator's system will provide tidal volume estimates within 15% of the respiratory monitor reference measurement, as well as respiratory rate estimates that closely match the respiratory monitor. The investigator's system employs a method that detects when the patient exhales and removes mask pressure during exhalation, and the investigators anticipate that this will result in improved comfort for the patient, as well as improved carbon dioxide monitoring accuracy, since removing flow during exhalation reduces dilution of the expired gas sample that is used for measuring exhaled carbon dioxide levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Have any respiratory or cardiovascular conditions
* i.e., cold, allergies, congestion, pneumonia, lung cancer, COPD, acute respiratory distress syndrome, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Tidal Volume Accuracy | During the intervention
  The mean and standard deviation of the percent difference in tidal volume measurement between our PAP system and the respiratory monitor

SECONDARY OUTCOMES:
Respiratory Rate | During the intervention
  The average respiratory rate reported by the respiratory monitor and rate reported by the PAP system for each volunteer will be compared. The average difference for each volunteer will be calculated, and a 95% confidence interval will be constructed, with the ideal mean difference being zero with low variance.
EtCO2 | During the intervention
  End-tidal carbon dioxide measurements at 10 cmH2O of mask pressure will be compared between when the system turned off flow during exhalation and when delivering flow throughout the entire breath. We anticipate that end-tidal CO2 levels will read lower when flow is delivered continuously during exhalation because of dilution of the expired gas, and this will be demonstrated by calculating the average difference in end-tidal CO2 between these two approaches.
Mask Pressure Control Accuracy | During the intervention
  The measured pressure in the mask compared to the set pressure in the 50 milliseconds immediately preceding inhalation will be assessed for evaluating pressure control. Average differences at each set pressure will be calculated. We anticipate these numbers to be less than 1 cmH2O.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Kuck, PhD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burk KM, Sakata DJ, Kuck K, Orr JA. Comparing Nasal End-Tidal Carbon Dioxide Measurement Variation and Agreement While Delivering Pulsed and Continuous Flow Oxygen in Volunteers and Patients. Anesth Analg. 2020 Mar;130(3):715-724. doi: 10.1213/ANE.0000000000004004. PMID 30633057
- [Background] Fogarty M, Orr JA, Sakata D, Brewer L, Johnson K, Fang JC, Kuck K. A comparison of ventilation with a non-invasive ventilator versus standard O2 with a nasal cannula for colonoscopy with moderate sedation using propofol. J Clin Monit Comput. 2020 Dec;34(6):1215-1221. doi: 10.1007/s10877-019-00426-5. Epub 2019 Nov 23. PMID 31760586